CLINICAL TRIAL: NCT04574700
Title: Effect of Knee Joint Mobilization on Hamstring Muscle Length
Brief Title: Mobilization Effect on Hamstring Length
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00688 Fareeha Sherazi
Record Dates: First submitted 2020-09-19; First posted 2020-10-05 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Mobilization; muscle length; knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Traction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- knee joint mobilization and traction (Experimental): Tibiofemoral, Tibiofibular joint anterioposterior mobilization, keltonborn knee traction Transcutaneous electrical nerve stimulation(TENS) and quadriceps strengthening
  Interventions: Other: knee joint mobilization and traction
- Post isometric relaxation (Active Comparator): Post isometric relaxation on hamstring, TENS and quadriceps strengthening.
  Interventions: Other: Post isometric relaxation

INTERVENTIONS:
Other: knee joint mobilization and traction — Grade 3 traction (Kaltenborn)from knee fully flexed to end of available Range of motion(ROM). Traction 30 sec, 10 sec rest period, 4reps, total 2 min of traction.3 sets for a total of 6 min of traction mobilization.Grade3 keltonborn tibiofemoral and tibiofibular anterior, posterior mobilization 3 sets10glides/set, 3 times/week on alternative days for 4 weeks.
  TENS for 20 mins in sitting and strengthening exercises i.e. Quadriceps Setting10 reps, air Cycling 2 min for a bout, straight leg raise (SLR) with weight , Full arc extension 10 reps of each exercise will be carried per session except for full-arc extension and air cycling. Air cycling cont. for 2 min for 1 bout of exercise. Measurement will be taken at base level, after first and last session. Treatment will be given for 3 times/week on alternative days for 4 weeks
  Arms: knee joint mobilization and traction
Other: Post isometric relaxation — Control group include Post isometric relaxation technique on hamstring muscle will be performed in supine lying, hip flexed to 90 degrees knee extended until the point of resistance 20% of maximum effort will be used by patient to create isometric contraction. Patient will be asked to breathe in and hold for 5 to 8 seconds and release both breath and effort then move to new barrier point and process was repeated three times per session
  TENS and strengthening exercises as mentioned above.
  This treatment regime will be given for 3 times/week on alternative days for 4 weeks.
  Arms: Post isometric relaxation

SUMMARY:
The aim of this research is to determine the effect of knee joint mobilization in patients with knee osteoarthritis having hamstring tightness. Tibiofemoral and tibiofibular joint mobilization and knee traction effect on hamstring muscle length and pain. A randomized controlled trial will be done at Benazir Bhutto Hospital Rawalpindi. The sample size is 44. The Participants are divided into two groups, 22 participants in experimental group and 22 in control group. The study duration is 6 months. Sampling technique applied is purposive non probability sampling technique, patients having Minimum 20% hamstring length shorting, NPRS more than 3,both gender of age 40-65,Pain more than 3 months and with mild to moderate knee OA are included. Tools used in this study are Numerical pain rating scale (NPRS), Goniometer and Western Ontario and McMaster Universities Arthritis Index (WOMAC) scale. Data analyzed through Statistical Package for the Social Science (SPSS)version 23.

DETAILED DESCRIPTION:
Knee Osteoarthritis is a type of joint disease or common rheumatologic disease that result from breakdown of joint cartilage and underlying bone which is characterized by pain, stiffness, and decreased range of motion. Knee OA is more important not only for its high prevalence rate compared with other types of OA but also for its presentation at earlier age groups particularly in younger age groups of obese women. Symptoms of knee OA progress slowly over years. The incidence of knee OA increases by age and further increase with longer lifetime and higher average weight of the population.

Symptoms of knee OA progress slowly over years. Pain and other symptoms of OA may have a profound effect on quality of life affecting both physical function and psychological parameters. Knee OA is not a localized disease of cartilage alone but is considered as a chronic disease of the whole joint, including articular cartilage, meniscus, ligament, and peri-articular muscle that may result from multiple pathophysiological mechanisms. It is painful and disabling disease that affects millions of patients.

Common symptoms are progressive knee stiffness, pain, difficulties in performing activities such as walking, stair climbing, squatting. Reduction in functional capacity associated with muscular imbalance of lower extremity with pain. Muscles act as brace for knee joint, quadriceps muscle weakness and hamstring inhibition effect this bracing. Muscle dysfunction may actually precede and accelerate the cartilage deterioration. Evidence showed muscle dysfunction is involved in pathogenesis of knee OA. Osteoarthritis (OA) is the most prevalent joint disease and a leading source of chronic pain and disability in the United States. Knee OA accounts for more than 80% of the disease's total burden and affects at least 19% of American adults aged 45 years and older.

Clinical strategies exist for treatment of knee osteoarthritis with aim to reduce symptoms like pain, delay disease progression i.e. pharmacological, physiotherapy and surgical strategies. Patients experience chronic pain that cause reduction in ability to use their joint. Due to prolong inactivity of joint to move through complete range cause muscle shortness along with capsule tightness that leads for further increasing pain and disability. Physical therapy interventions are first line of choice for the treatment of knee OA. Treatment varieties i.e. modalities, therapeutic exercises, manual therapy along with neuromuscular training to improve mechanical environment of knee joint

It is indicated at least 15-30 degree loss of active knee extension with 90 degree of hip ﬂexion account as hamstring shortening. Hamstring muscle tightness and poor flexibility is associated with knee OA. Hamstring flexibility is higher in healthy individual as compared to subjects with knee OA.A statistically significant relationship was found between hamstring tightness and proximal tibiofibular joint grade of arthritis (χ2 test, p=0.004) Recent study reported 97.6% of middle aged men with hamstring muscle tightness Hamstring flexibility is greater in females than males. Research showed that ischio-tibial flexibility reduce pain stiffness and significant functional limitation in knee OA. Joint mobilizations are most widely used in treatment of knee OA having various neuro-physiological effects including decrease in pain, stiffness, activation and inhibition of muscles.The muscular system reflects sensorimotor system it receives information from musculoskeletal and central nervous systems. Changes occur in tone within the muscle are the first responses to nociception by the sensorimotor system. Many studies reported effect of joint pathology on muscle tone for example the presence of knee effusion causes reflex inhibition of the vastus-medialis and multifidus has been shown to atrophy in patients with chronic low back pain. In this study we aim to increase hamstring muscle length through activation of mechanoreceptors by mobilizations.

There is no study conducted yet to determine effect of joint mobilization on adjacent muscle length other than soft tissue techniques which are mainly stretches.

Literature review: randomized control trail (2019) conducted for comparing effectiveness on Proprioceptive Neuromuscular Facilitation(PNF) stretching verses static stretching on hamstring flexibility in knee OA patients showed PNF stretching was better in outcome measures

A study compared static verses intermittent stretching for increase of hamstring muscle length concluded that intermittent stretching is more effective for hamstring flexibility.

A pre-post study (2019) find out effect of unilateral posteroanterior mobilization(UPA) on lumbar spine observed in his study that UPA lumbar mobilizations increased lumbar Range of Motion and hamstring extensibility by a moderate magnitude and this effect remained for 10-15 minutes post treatment.

Study reported Joint manipulations reduce nociceptor stimulus, depress responsiveness of alpha motor neurons causing changes in muscle tone.

Study on active stretching and passive mobilization of cervical spine for neck pain concluded there was increase range of motion in both groups.

comparing Muscle Energy Technique(MET) with conventional treatment for hamstring flexibility in knee OA patients reported that MET was better than conventional treatment.

A randomized control trail(2014)compared immediate effects of neurodynamics slider technique verses static stretch concluded neurodynamics slider technique is more effective for improving hamstring flexibility.

Therapeutic effect of joint mobilization that joint mobilization may promote muscles relaxation thereby increasing joint range of motion

Joint mobilization and traction allows for selective stretching of selected tissue and can be expected to change both elastic and plastic component of stiffness. The intermittent compression and distraction of joint distribute fluid into soft tissue decreasing spasm allowing for easier movement and increase range of motion.

Joint mobilization cause stimulation of Golgi tendon organ activity, and reflex inhibition of the muscle at the end of the passive joint mobilization.

A study concluded that joint mobilization decreases muscle activity, reducing muscle concentric activation, pain, and muscle tension in periarticular-tissue

ELIGIBILITY:
Inclusion Criteria:

* Minimum 20% length shorting
* NPRS more than 3
* Gender include male and female
* Age 40-65
* Pain more than 3 months.
* Patients with mild to moderate knee OA (primary and secondary) grade 1and 2 Kellgren and Lawrence classification system based on plain x-rays taken in supine lying position. They should satisfy the American College of Rheumatology Criteria for clinical classification of knee OA.

Hamstring shortness screening criteria: following tests should be positive for participants to enroll in this study

* Active knee extension test
* 90-90 test
* Sit and reach test

Exclusion Criteria:

* Co morbidities (i.e. Systematic diseases)
* Patient on long-term Medications i.e. corticosteroid
* Patient with Spinal Surgery
* Recent trauma
* Hamstring contracture.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Hamstring length: (Active Knee Extension Test) | 12th day
  Changes from the baseline to 12th day, this test is for to check hamstring flexibility, Patient position is in supine and effected leg is in 90 degree hip flexion. Patient is asked to extend the knee. Cutoff value for the Active knee extension test is 160.Normal individual presents with>160 or equal to160 (=160) and angle <160 considered hamstring tightness.

SECONDARY OUTCOMES:
Numeric Pain rating scale (NPRS) | 12th day
  Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain
WOMAC Scale | 12th day
  Changes from baseline WOMAC scale, it's a scale to evaluate the condition of patients with osteoarthritis of the knee, consisting of 24 items divided into 3 subscales including pain (5 items), stiffness (2 items), and physical functioning (17 items) of the joints.There are 5 responses to each question having a score assigned to it like None=0,slight=1,moderate=2,severe=3,extreme=4.scoring of this scale is done by sum up of all the points,minimum possible score is 0 while maximum possible score is 96.Higher number represents higher levels of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Saira Waqqar, PPDPT,MHPE, Principal Investigator — Riphah international universty
Locations (1):
- Riphah International University Islamabad, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hides JA, Stokes MJ, Saide M, Jull GA, Cooper DH. Evidence of lumbar multifidus muscle wasting ipsilateral to symptoms in patients with acute/subacute low back pain. Spine (Phila Pa 1976). 1994 Jan 15;19(2):165-72. doi: 10.1097/00007632-199401001-00009. PMID 8153825
- [Background] Chen JG CE, Kim MK. Immediate Effect of Intermittent Versus Continuous Hamstring Static Stretching on the Muscle Tone and Range of Motion. 대한물리의학회지. 2019(14(4)):19-27
- [Background] N S. A comparative study on the effectiveness of PNF stretching versus static stretching on Pain and Hamstring flexibility in osteoarthritis knee patients. International Journal of Research in Pharmaceutical Sciences. 2019 Jul 12;10(3):1789-94
- [Background] Chesterton P, Evans W, Livadas N, McLaren SJ. Time-course changes associated with PA lumbar mobilizations on lumbar and hamstring range of motion: a randomized controlled crossover trial. J Man Manip Ther. 2019 May;27(2):73-82. doi: 10.1080/10669817.2018.1542558. Epub 2018 Nov 13. PMID 30935338
- [Background] Kim S-H, Choi J-H, Lee K-W. Immediate effects of active stretching versus passive mobilization of the upper cervical spine on patients with neck pain and ROM. Korean Society of Physical Medicine. 2016;11(4):27-32
- [Background] Choksi P TK. To Study the Efficacy of Muscle Energy Technique on Muscle Strength and Flexibility in Patients with Knee Osteoarthritis. . Indian Journal of Physiotherapy and Occupational Therapy-An International Journal. 2016;10((3)):40-5
- [Background] Castellote-Caballero Y, Valenza MC, Puentedura EJ, Fernandez-de-Las-Penas C, Alburquerque-Sendin F. Immediate Effects of Neurodynamic Sliding versus Muscle Stretching on Hamstring Flexibility in Subjects with Short Hamstring Syndrome. J Sports Med (Hindawi Publ Corp). 2014;2014:127471. doi: 10.1155/2014/127471. Epub 2014 Apr 15. PMID 26464889
- [Background] Kahanov L, Kato M. Therapeutic effect of joint mobilization: joint mechanoreceptors and nociceptors. Athletic Therapy Today. 2007;12(4):28-31
- [Background] Randall T, Portney L, Harris BA. Effects of joint mobilization on joint stiffness and active motion of the metacarpal-phalangeal joint. J Orthop Sports Phys Ther. 1992;16(1):30-6. doi: 10.2519/jospt.1992.16.1.30. PMID 18796775
- [Background] Zusman M. Spinal manipulative therapy: review of some proposed mechanisms, and a new hypothesis. Aust J Physiother. 1986;32(2):89-99. doi: 10.1016/S0004-9514(14)60645-0. PMID 25026443
- [Background] Lundberg A, Malmgren K, Schomburg ED. Role of joint afferents in motor control exemplified by effects on reflex pathways from Ib afferents. J Physiol. 1978 Nov;284:327-43. doi: 10.1113/jphysiol.1978.sp012543. PMID 215758